CLINICAL TRIAL: NCT04676009
Title: Feasibility of an Acute Physical Exercise Before Immunotherapy and Chemotherapy Infusion for Metastatic Non-small-cell Lung Cancer Patients: Protocol ERICA Study
Brief Title: Feasibility of an Acute Physical Exercise Before Treatment Infusion for Metastatic Lung Cancer Patients
Acronym: ERICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Claude Bernard University (Other); Lyon Cancer Research Centre (Unknown); Hospices Civils de Lyon (Other); Inter-university Laboratory of Human Movement Biology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERICA; ET20000185 (Other: Sponsor's ID)
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lung Cancer; Lung Neoplasm; Metastasis; Acute exercise; Immunotherapy; Connected devices
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise arm : (Experimental): Patient randomized to the Exercise arm will receive physical activity recommendations at inclusion and nutritional assessment will be carried out during the first and last treatment cure. Patients will receive an acute physical exercise just before immunotherapy and chemotherapy infusion.They will have a home walking program and will have to wear an activity tracker during the 3 months of intervention.
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place before exercise (1), after exercise (2) and 12 hours after the start of treatment (3).
  Interventions: Other: Exercise arm :
- Control arm (No Intervention): Patients will receive physical activity recommendations at inclusion and a nutritional assessment will be carried out during the first and last treatment cure. They will receive the usual care and standard treatment protocol (immunotherapy and chemotherapy).
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment (3).

INTERVENTIONS:
Other: Exercise arm : — Patients will receive physical activity recommendations at inclusion.
  At each treatment cure, patients will receive pre-exercise nutritional recommendations and an acute physical exercise prior to immunotherapy and chemotherapy. The acute physical exercise will last 35 minutes and will be intermittent and individualized based on the results obtained by the patient during an endurance test on a ergocyle performed prior to treatment.
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place before exercise (1), after exercise (2) and 12 hours after the start of treatment (3).
  A nutritional assessment will be carried out during the first and last treatment cure.
  They will also benefit a home walking program. These patients will have to wear an activity tracker tracker during all intervention (3 months).
  They will have a phone follow-up every 10 days (± 3 days) after each treatment cure for the study duration.
  Arms: Exercise arm :

SUMMARY:
Because of metastatic Non-Small Cell Lung Cancer (mNSCLC) and its treatments, patients suffer from numerous symptoms such as dyspnea, muscle atrophy, pain, fatigue, loss of appetite, altered physical condition and lung function, which may further impair the patient's overall condition. Nevertheless, it has been suggested that physical exercise could improve response to treatment at the clinical level due to its known effects on the immune system. Moreover, preclinical studies have shown that exercise performed during chemotherapy administration could result in physiological benefits such as improved intra-tumoral infusion and drug delivery. The ERICA study aims to assess the feasibility of an acute physical exercise immediately before immunotherapy and chemotherapy administration in patients with mNSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years old,
* Having a newly metastatic non-small-cell lung cancer (NSCLC) without an EGFR/ALK alteration diagnosis,
* Being scheduled to receive a 1st line intravenous chemotherapy (Cisplatin and Pemetrexed or Carboplatin and Pemetrexed or Taxol and Carboplatin), and immunotherapy (monoclonal anti-PD-1 and anti-PD-L1 antibodies : Pembrolizumab) treatment NB : patients who have previously received one or more treatments other than chemotherapy (e.g. targeted therapy) and must start their first chemotherapy are eligible,
* Treated in Centre Leon Berard,
* Having an Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2,
* Being voluntary and available to get involved throughout the study duration,
* Being able to engage in Physical Activity with a medical certificate attested by one of the investigators clinical oncologist or the referring oncologist,
* Affiliated with a social security scheme,
* Having dated and signed an informed consent.
* Able to read, write and understand French

Exclusion Criteria:

* Patient with unstable bone metastases or unconsolidated pathologic fractures, Having a central nervous system impairment with neurological disorder avoids the physical exercise practice on a cycle ergometry,
* Personal history or co-existence of another primary cancer (except of in situ cancer regardless of the site and/or basal cell skin cancer and/or cancer in complete remission for more than 5 years),
* Having severe undernutrition defined according to the Haute Autorité de Santé (i.e. , for an adult aged ≥18 years and < 70 : BIM ≤ 17 or weight loss ≥ 10% in 1 month or ≥15% in 6 months or ≥ 15% compared to the usual weight before the disease diagnosis or albuminemia < 30 g/l ; for an adult aged ≥70 years : BIM < 18 or weight loss ≥ 10% in 1 month or ≥15% in 6 months or an albuminemia < 30 g/l),
* Having a severe amenia (hemoglobin ≤ 8 g/dl) during the 30 last days prior inclusion,
* Presenting cardiovascular history or any cardiovascular risk: chronic coronary (or poorly balanced), artery disease, cardiac arrhythmia, symptomatic heart disease, uncontrolled or untreated hypertension, heart attack diagnosed within the last 6 months, coronary angioplasty with or without stent less than 6 months old, coronary artery bypass surgery less than 12 months old, history of poorly balanced type 2 diabetes,
* In case of diabetes: Glycated hemoglobin (HbA1c) > 7% (in the last 3 months),
* Stage IV Chronic Obstructive Pulmonary Disease (FEV1 < 30%),
* Patient with a contraindication to the proposed physical exercise in the study (orthopedic disorder likely to impede walking and pedaling such as disabling coxarthrosis or gonarthrosis, operated or not),
* Already included in a PA study,
* Cannot be followed for medical, social, family, geographical or psychological reasons, for the duration of the intervention (3 months) and then for the duration of the post-intervention follow-up (3 months),
* Patient under legal protection measure (under guardianship, curatorship, safeguard of justice),
* Deprived of liberty by judicial or administrative decision,
* Pregnant patient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Investigate the feasibility of an acute physical exercise during the immunotherapy/chemotherapy preinfusion | 3 months
  Ratio of the number of acute physical exercise sessions immunotherapy/chemotherapy preinfusion performed by"exercise" group patient / number of acute physical exercise sessions planned

SECONDARY OUTCOMES:
Investigate the physical activity fitness (sub-maximum endurance test) | Baseline, 3 months
  Sub-maximum endurance test on an ergocycle
Investigate the lower strength muscular function change | Baseline, 3 months, 6 months
  Maximum isometric force of the knee extensors
Investigate the maximum isometric upper limb strength change | Baseline, 3 months, 6 months
  Hand dynamometer
Investigate the Physical Activity level change | Baseline, 3 months, 6 months
  The PA level will be measured by the Godin Leisure-Time Physical Activity Questionnaire (GLTAPQ). The GLTAPQ is a 4-item self-administered questionnaire with the first three questions designed to obtain information on the number of times an individual engages in light, moderate and intense "leisure-time PA" periods of at least 15 minutes during a typical week. The scoring of the GSLTPAQ is the "LSI" (Leisure Score Index) is obtained using the following formula: (light PA frequency × 3) + (moderate PA frequency × 5) + (vigorous PA frequency × 9). People with a moderate to high LSI ≥ 24 are classified as active, while people reporting a moderate to high LSI ≤ 23 are classified as insufficiently active (estimated energy expenditure < 14 Kcal/kg/week).
Investigate the patient anthropometrics change | Baseline, 3 months, 6 months
  Weight in kilograms
Investigate the patient anthropometrics change | Baseline, 3 months, 6 months
  Hip circumference in centimeters
Investigate the patient anthropometrics change | Baseline, 3 months, 6 months
  Waist circumference in centimeters
Investigate the patient anthropometrics change | Baseline, 3 months, 6 months
  BMI (weight/height²)
Investigate the patient health-related quality of life change | Baseline, 3 months, 6 months
  Quality of life will be measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality Of Life Questionnaire (QLQ-C30). Quality of life specific to lung cancer will be assessed by the 13-item module: The Quality Of Life Questionnaire - Lung Cancer 13 (QLQ-LC13). The QLQ-LC13 self-questionnaire is an additional measure of the symptoms and side effects experienced by lung cancer patients who receive non-surgical treatment.
Investigate the patient health-related quality of life specific to lung cancer change | Baseline, 3 months, 6 months
  Quality of life specific to lung cancer will be assessed by the 13-item module: The Quality Of Life Questionnaire - Lung Cancer 13 (QLQ-LC13). The QLQ-LC13 self-questionnaire is an additional measure of the symptoms and side effects experienced by lung cancer patients who receive non-surgical treatment.
Investigate the fatigue change | Baseline, 3 months, 6 months
  Fatigue will be assessed by the EORTC-QLQ module measuring cancer-related fatigue (EORTC QLQ-FA12). This self-questionnaire includes 12 items that assess physical, cognitive and emotional fatigue related to cancer. Participants will respond on a Likert scale ranging from "not at all" to "a lot". All scores will be transformed into a scale from 0 to 100, with a higher score indicating a higher degree of fatigue.
Investigate the sleep quality change | Baseline, 3 months, 6 months
  The perceived quality of sleep is assessed by the Insomnia Severity Index (ISI) which measures the severity of insomnia. The questionnaire consists of 7 items rated on a 5-point scale ranging from 0 ("none") to 4 ("very severe"). This self-questionnaire makes it possible to evaluate the severity of the patient's sleep difficulties (initial, maintenance, morning insomnia), the degree of sleep dissatisfaction, the level of interference with daily functioning, the degree of appearance of sleep difficulties and the level of anxiety related to insomnia. The total score of the items varies between 0 and 28. A high score indicates greater sleep difficulties.
Investigate the impact of social vulnerability | Baseline
  Social vulnerability will be assessed by the EPICES score (Evaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé). By adding up the points of the 11 binary questions ("Yes"/"No") of the self-questionnaire we obtain the so-called EPICES score. This quantitative score varies from 0 "no precariousness" to 100 "highest precariousness".
Investigate the muscle mass and sarcopenia | Baseline, 3 months, 6 months
  CT scans
Investigate the immune biomarkers change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
  The following immune biomarkers will be assay : Natural Killer cells, B lymphocytes, T lymphocytes, monocytes, sub-populations of dendritic cells on frozen PBMC
Investigate the Activin change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the TNF-alpha change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the IL-1béta change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the IL-6 change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Follistatin (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the GDF5 (BMP14) (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the GDF15 (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the IL-10 (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the IL-15 (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the NH3 (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Aminogramme (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the CRP (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the IFN-gamma change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Cortisol change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Myostatin change (inflammation biomarkers) | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Advanced oxidation protein products (AOPP) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the Superoxide dismutase (SOD) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the catalase (CAT) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the malondialdehyde (MDA) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
  The following biomarkers will be assay : Advanced oxidation protein products (AOPP), malondialdehyde (MDA), Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX), Xanthine oxidase (XO), and Myeloperoxidase (MPO).
Investigate the glutathione peroxidase (GPX) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
  The following biomarkers will be assay : Advanced oxidation protein products (AOPP), malondialdehyde (MDA), Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX), Xanthine oxidase (XO), and Myeloperoxidase (MPO).
Investigate the Xanthine Myeloperoxidase (MPO) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
  The following biomarkers will be assay : Advanced oxidation protein products (AOPP), malondialdehyde (MDA), Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX), Xanthine oxidase (XO), and Myeloperoxidase (MPO).
Investigate the Xanthine oxidase (XO) change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
  The following biomarkers will be assay : Advanced oxidation protein products (AOPP), malondialdehyde (MDA), Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase (GPX), Xanthine oxidase (XO), and Myeloperoxidase (MPO).
Proportion of patients who have severe toxicity (grade >2) | Up to 3 months
  Occurence of severe toxicity (grade > 2) according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE). Number of delayed or cancelled treatment sessions and relative dose-intensity (RDI) for patients with grade ≥ 3 chemotherapy-related toxicities, calculated as the ratio of the "delivered" dose-intensity to the "expected" dose-intensity.
Progression free survival | 6 months
  Period from the date of randomization to the date of event defined as disease progression or death from any cause
Acceptability of the study | 3 months
  Ratio of the number of patients included / number of eligible patients
Tracker activity acceptability | 3 months
  Number of days the activity tracker is worn / number of days in the programme
Safety of the intervention | 3 months
  Number, type and timing of adverse events due to program
Adherence of the intervention | 3 months and 6 months
  number of steps at home realized / number of steps at home prescribed (only in the intervention arm)
Investigate the Physical Activity level change | Baseline, 3 months and 6 months
  Daily number of step prescription (only in the intervention arm)
Investigate the glucose change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the insulin change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the lactat change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the PCR change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).
Investigate the HIF-1 change | Baseline and 3 months
  3 blood sampling times (2 EDTAsx10 mL) will be specially added to the study and will take place: for the exercise group: before exercise (1), after exercise (2) and 12 hours after the start of treatment (3); and for the control group: 40 min before the administration of treatments (1), just before the administration of treatments (2) and 12 hours after the start of treatment(3).

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Pérol, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gouez M, Perol O, Perol M, Caux C, Menetrier-Caux C, Villard M, Walzer T, Delrieu L, Saintigny P, Marijnen P, Pialoux V, Fervers B. Effect of acute aerobic exercise before immunotherapy and chemotherapy infusion in patients with metastatic non-small-cell lung cancer: protocol for the ERICA feasibility trial. BMJ Open. 2022 Apr 7;12(4):e056819. doi: 10.1136/bmjopen-2021-056819. PMID 35393316